CLINICAL TRIAL: NCT06722261
Title: Single Case Research Design: Deaf Children's Language Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 478857; R21DC021024 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Language Development
Keywords: Sign Language; Deaf; Intervention
MeSH Terms: conditions — Sign Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Case Research Design: Phase 1 (Experimental): A randomized selection method will be employed to select deaf children to participate in single case research. Two children will be selected from each age group between 5 and 10, making a total of eight students. Their language skills will be closely monitored and evaluated over the course of the year. Following the noncurrent multiple baseline design, in succession across 8 child participants in 4 classes, 2 Phase 1 participants in a class will begin receiving SISI while other children remain in the baseline for 3 to 9 weeks.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Phase 2 (Experimental): A randomized selection method will be employed to select deaf children to participate in single case research. Two children will be selected from each age group between 5 and 10, making a total of eight students. Their language skills will be closely monitored and evaluated over the course of the year. Following the noncurrent multiple baseline design, in succession across 8 child participants in 4 classes, three weeks after Phase 1 participants have begun SISI, Phase 2 participants in a class will begin receiving SISI while other children remain in the baseline.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Phase 3 (Experimental): A randomized selection method will be employed to select deaf children to participate in single case research. Two children will be selected from each age group between 5 and 10, making a total of eight students. Their language skills will be closely monitored and evaluated over the course of the year. Following the noncurrent multiple baseline design, in succession across 8 child participants in 4 classes, 2 SCRD participants in a class will begin receiving SISI while other children remain in the baseline for 3 weeks.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Phase 4 (Experimental): A randomized selection method will be employed to select deaf children to participate in single case research. Two children will be selected from each age group between 5 and 10, making a total of eight students. Their language skills will be closely monitored and evaluated over the course of the year. Following the noncurrent multiple baseline design, in succession across 8 child participants in 4 classes, 2 SCRD participants in a class will begin receiving SISI while other children remain in the baseline for 3 weeks.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction

INTERVENTIONS:
Behavioral: Strategic and Interactive Signing Instruction — Evidence-based instructional methods, grounded in cognitive, sociocultural, and linguistic theories, are applied to interventions that support sign language development in deaf children.

SUMMARY:
Eight deaf children in kindergarten to 3rd grade classes will be randomly selected for single case research. Their language skills will be monitored and assessed daily. Using a noncurrent multiple baseline design (Single Case Research Design or SCRD), Strategic and Interactive Signing Instruction (SISI) will be administered to two children in each of four classes.

DETAILED DESCRIPTION:
A randomized selection method will be employed to select deaf children to participate in single case research. Two children will be selected from each age group between 5 and 10, making a total of eight students. Their language skills will be closely monitored and evaluated over the course of the year. Following the noncurrent multiple baseline design, in succession across 8 child participants in 4 classes, 2 SCRD participants in a class will begin receiving SISI while other children remain in the baseline for 3 weeks. Brainstorming occurs on Monday and the final sign language composition is shared on Friday. At the end of each day's intervention, child participants will independently narrate their expressed message recorded on videos. A score of 1 (applied correctly), 0.5 (applied but incorrectly), or 0 (omitted) will be given to their inclusion of target sign language skills, which is converted into percentages. If a child receives 100% on their target SL skill for 3 consecutive days (3 data points), Teacher 1 will select a new sign language skill to target. If the child receives 0% or 50% on their target sign language skill, Teacher 1 continues to focus on the same sign language skill.

ELIGIBILITY:
Inclusion Criteria:

* Deaf children in kindergarten to 3rd grade class in a school for the deaf

Exclusion Criteria:

* Non-deaf children

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Sign Language Skills | From enrollment to the end of treatment 9 academic months later.
  Deaf children's development of target sign language skills will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Under a data-sharing agreement that is in compliance with the internal policy at UTK, non-identifying data can be shared with other researchers for a minimum of 10 years on the University of Tennessee Research and Creative Exchange (TRACE). The raw data consists of videos of teachers, which will not be shared to maintain confidentiality. The processed data will be in the form of percentages for individual teachers across an academic year documented in a .csv file (Excel). Center for Open Science Foundation (OSF) is a free and open source project management tool that supports researchers throughout their entire project lifecycle. OSF also allows people to locate this data through project names, author names, and study keywords.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: December, 2026 to December, 2036
Access Criteria: Researchers may contact the principal investigator for additional supporting information not available on OSF.